CLINICAL TRIAL: NCT04637529
Title: National, Multicentre, Randomized, Double-blind, Double-dummy Phase II Clinical Trial to Evaluate the Efficacy and Safety of S (+) - Ibuprofen for Pain Control in Individuals With Osteoarthritis
Brief Title: Efficacy and Safety of S (+) - Ibuprofen in Osteoarthritis Pain
Acronym: APS003/2020
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APS003/2020
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis
Keywords: Nonsteroidal anti-inflammatory; Pain; Ibuprofen; Inflammation; Anti-inflammatory; Pain control; Osteoarthritis; Pain relief; Enzyme Inhibitors
MeSH Terms: conditions — Osteoarthritis; Pain; Inflammation; Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S (+) - Ibuprofen (Experimental): S (+) - Ibuprofen (1 coated tablet) + placebo of Ibuvix® - ibuprofen (1 coated tablet) Every 6 hours for 28 days.
  Interventions: Drug: S (+) - Ibuprofen
- Ibuvix® - ibuprofen (Active Comparator): Ibuvix® - ibuprofen (1 coated tablet) + placebo of S (+) - Ibuprofen (1 coated tablet) Every 6 hours for 28 days.
  Interventions: Drug: Ibuvix® - ibuprofen

INTERVENTIONS:
Drug: S (+) - Ibuprofen — S (+) - Ibuprofen + placebo of Ibuvix®
  Arms: S (+) - Ibuprofen
Drug: Ibuvix® - ibuprofen — Ibuvix® + placebo of S(+) - Ibuprofen
  Arms: Ibuvix® - ibuprofen

SUMMARY:
The purpose of this study is to evaluate the efficacy of S (+) - ibuprofen compared to an active treatment for pain control in individuals diagnosed with osteoarthritis.

ELIGIBILITY:
Main Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Patients aged from 18 to 75 with a diagnosis of knee and/or hip osteoarthritis according to American College of Rheumatology (ACR) criteria.

Main Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* Previous history of alcohol or drugs abuse diagnosed by DSM-V;
* Current or previous history (less than 12 months) of smoking;
* Have clinically relevant abnormal laboratory results according to medical evaluation;
* Women who are pregnant, lactating, or positive for β - hCG urine test;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mean reduction of pain measured by the WOMAC Osteoarthritis Index (pain) | Baseline (day 0) and Week 4 (day 28)

SECONDARY OUTCOMES:
Patient Global Impression of Improvement-I (PGI-I) | Week 4 (day 28)
Proportion of participants among the groups to discontinue the trial due to treatment non-tolerability | From Baseline (day 0) to Week 4 (day 28)

CONTACTS AND LOCATIONS:
Locations (1):
- Apsen Farmacêutica S.A., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No